CLINICAL TRIAL: NCT00472485
Title: Study of Eye Movement Testing and Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00H0185
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Saccadic Eye Movement Deficiency; Oculomotor Deficiency; Oculomotor Dysfunction

INTERVENTIONS:
Procedure: eye movement therapy

SUMMARY:
The purpose of this study is to determine the ability of several eye movement monitors, used in clinical practice, to identify children with poor reading eye movements. A second purpose of the study is to evaluate the effectiveness of eye movement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8 to 13 with saccadic eye movement deficit

Exclusion Criteria:

* Previous saccadic eye movement therapy

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Marjean Kulp, OD, MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States